CLINICAL TRIAL: NCT01517451
Title: Stereotactic Body Radiation Therapy and Short-Term Androgen Ablation for Intermediate-Risk, Localized, Adenocarcinoma of the Prostate
Brief Title: Radiation and Androgen Ablation for Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11157; NA_00067963 (Other: JHMIRB)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma of the Prostate
MeSH Terms: interventions — Radiotherapy; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation with Androgen Deprivation Therapy (ADT) (Experimental): This will be a Phase I/II study evaluating the effectiveness and toxicity of a combined regimen of 7.25 Gy every other day fractions to a total dose of 36.25 Gy (total of 5 fractions) with androgen deprivation therapy (ADT) for 4 months total, greater than or equal to 1 month prior to SBRT (stereotactic body radiation therapy). This choice of daily dose is based on the prior published experience showing safety and efficacy of hypofractionated regimens.
  Interventions: Radiation: Radiation Therapy; Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Radiation: Radiation Therapy — 7.25 Gy every other day fractions to a total dose of 36.25 Gy (total of 5 fractions)
Drug: Androgen Deprivation Therapy (ADT) — Androgen deprivation therapy (ADT) for 4 months total, greater than or equal to 1 month prior to SBRT.

SUMMARY:
A study to see how effective and tolerable radiation therapy along with androgen deprivation therapy is in treating prostate cancer.

DETAILED DESCRIPTION:
This will be a Phase I/II study evaluating the effectiveness and toxicity of a combined regimen of 7.25 Gy every other day fractions to a total dose of 36.25 Gy (total of 5 fractions) with androgen deprivation therapy (ADT) for 4 months total.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally confined adenocarcinoma of the prostate
* Patient must fit D'Amico intermediate risk criteria by clinical stage (T2b-T2c), PSA (prostatic specific antigen) (10-20 ng/mL), and/or Gleason score (Gleason 7).
* The patient has decided to undergo external beam radiation as treatment choice for his prostate cancer.
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Stage T3-4 disease.
* Gleason 8 or higher score.
* PSA > 20 ng/ml.
* IPSS (International Prostate Symptom Score) > 15
* Clinical or Pathological Lymph node involvement (N1).
* Evidence of distant metastases (M1).
* Radical surgery for carcinoma of the prostate.
* Previous Chemotherapy, unless intervention was greater than 5 years from beginning treatment for current prostate cancer.
* Previous pelvic radiation therapy.
* Previous or concurrent cancers other than basal or squamous cell skin cancers or superficial bladder cancer unless disease free for at least 5 years.
* History of inflammatory bowel disease.
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow up.
* Myocardial infarction or cerebrovascular accident within one year from consultation, or other major vascular risk factor which would prevent a patient from receiving appropriate androgen deprivation therapy.11
* Liver function tests (LFTs) greater than twice the upper limit of normal.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Song, M.D., Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Started | 45
Completed | 44
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 65 [56 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Failure Free-rate (BFFR) Associated With the Combined Hypofractionated Dose Regimen and Androgen Deprivation Therapy (ADT).
Description: To assess 5-year biochemical failure free rate (BFFR) associated with image-guided radiation therapy in doses of 7.25 Gy every other day to a total dose of 36.25 Gy (5 fractions) along with 4 months of androgen deprivation therapy (ADT) neoadjuvantly and concurrently. BFFR is defined as binary indicator whether PSA has increased by 2 ng/ml or more above the nadir PSA any time before the end of 5 years as the number of events.
Time Frame: From consent up to 5 years post treatment completion
Measure: Number; unit: progression events
Groups:
- Radiation With Androgen Deprivation Therapy (ADT): Patients receiving combined regimen of radiation therapy 7.25 Gy every other day fractions to a total dose of 36.25 Gy (total of 5 fractions) with androgen deprivation therapy (ADT) for 4 months total, greater than or equal to 1 month prior to SBRT (stereotactic body radiation therapy).
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
progression events | 0

2. Secondary Outcome: Toxicity as Assessed as Incidence of Grade 3 or Greater Gastrointestinal (GI) and Genitourinary (GU) Adverse Events
Description: Incidence of grade 3 or greater GU (genitourinary) and GI (gastrointestinal) toxicity with image-guided radiation therapy in doses of 7.25 Gy every other day to a total dose of 36.25 Gy (5 fractions) along with 4 months of androgen deprivation therapy (ADT) neoadjuvantly and concurrently.
Time Frame: Consent to up to 5 years of follow-up or biochemical failure.
Measure: Number; unit: events
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 45
events
  GU | 4
  GI | 0

3. Secondary Outcome: Overall Survival Rate
Description: Assess clinical control rate by measuring the Overall Survival (OS) which is defined as the percentage of participants who completed the study that lived from time of treatment until death from any cause.
Time Frame: Start of treatment up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
Participants | 44

4. Secondary Outcome: Number of Patients Who Completed Blood Collection of Whole Blood for Future Research
Description: Biomarker studies. Number of patients who completed blood collection of whole blood for future research.
Time Frame: Up to 2 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
Participants | 10

5. Secondary Outcome: Self-reported Patient Quality of Life Data Using the International Prostate Symptom Score (IPSS).
Description: The International Prostate Symptom Score (IPSS) is a useful subjective assessment tool for Benign prostatic hyperplasia (BPH) patients; it is a modification of the American Urological Association (AUA) Symptom Index. The questionnaire assesses degree of Lower Urinary Tract Symptoms (LUTS) and quality of life. Patients can fill out the IPSS form before examinations, but minimal interference from health care providers must be ensured. Total score range 0-35; A score of 7 or less is mildly symptomatic, 8 to 19 is moderately symptomatic, and 20 to 35 is severely symptomatic.
Time Frame: Measured at baseline and at 3, 12, 24 and 36 months post treatment
Population: Patients with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
score on a scale
  Baseline: number analyzed (Participants) | 22
  Baseline | 7.32 (5.49)
  3 month Follow-up: number analyzed (Participants) | 28
  3 month Follow-up | 7.79 (5.77)
  12 month Follow-up: number analyzed (Participants) | 25
  12 month Follow-up | 7.91 (5.66)
  24 month Follow-up: number analyzed (Participants) | 1
  24 month Follow-up | 2.00 (NA) — Only one patient completed the IPSS assessment therefore a standard deviation cannot be calculated.
  36 month Follow-up: number analyzed (Participants) | 29
  36 month Follow-up | 6.82 (4.88)

6. Secondary Outcome: Patient Reported Sexual Health Inventory for Men (SHIM), a Self-reported Quality of Life Assessment
Description: The SHIM serves several key functions within clinical and research settings. Its core purpose involves screening for and evaluating the severity of erectile dysfunction (ED). Total score range 5 to 25; higher scores indicate better erectile function. A total score of 21 or less indicates erectile dysfunction. 22-25: No erectile dysfunction, 17-21: Mild ED, 12-16: Mild-to-moderate ED, 8-11: Moderate ED, 5-7: Severe ED.
Time Frame: Baseline and at 3,12, 24 and 36 months follow-up
Population: Patients with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
score on a scale
  Baseline SHIM: number analyzed (Participants) | 22
  Baseline SHIM | 15.3 (8.96)
  3 months: number analyzed (Participants) | 28
  3 months | 6.14 (8.99)
  12 months: number analyzed (Participants) | 25
  12 months | 7.16 (8.66)
  24 months: number analyzed (Participants) | 1
  24 months | 25.0 (NA) — [1] NA Explanation: Only one patient completed the SHIM assessment therefore a standard deviation cannot be calculated.
  36 months: number analyzed (Participants) | 29
  36 months | 6.79 (8.08)

7. Secondary Outcome: The Expanded Prostate Cancer Index Composite 26 (EPIC). Self-reported Quality of Life Assessment of Sexual Health
Description: The EPIC-26 (Expanded Prostate Cancer Index Composite-Short Form) is a validated questionnaire for measuring sexual health related quality of life. Scores range from 1 to 100, with higher scores being better score.
Time Frame: 3,12, 24 and 36 months follow-up
Population: At each timepoint the number of participants varies based on patient data collected for the EPIC assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 44
score on a scale
  3 months: number analyzed (Participants) | 28
  3 months | 34.7 (46.5)
  12 months: number analyzed (Participants) | 25
  12 months | 38.2 (34.3)
  24 months: number analyzed (Participants) | 1
  24 months | 100 (NA) — [1] NA Explanation: Only one patient completed the EPIC assessment therefore a standard deviation cannot be calculated.
  36 months: number analyzed (Participants) | 29
  36 months | 39.8 (27.6)

ADVERSE EVENTS:
Time Frame: From enrollment up to 5 years
Arm/Group | Radiation With Androgen Deprivation Therapy (ADT)
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation With Androgen Deprivation Therapy (ADT) (N=45)
Skin Infection (Infections and infestations) | 1 (1) — Pt. missed 4 year f/u due to 3-day hospitalization for cellulitis and continued outpatient IV abx for 28 days completed 2/29/2020. Also reported hyperglycemia Grade 4, also documented. History of DM on insulin with Charcot foot and severe neuropathy.
Syncope (Nervous system disorders) | 1 — The patient had a syncopal episode while working out at the gym. Patient was taken by ambulance to the Sibley ED, where he was evaluated for 2 hours and given IV fluids. The event most likely caused by dehydration. Was referred to cardiology.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation With Androgen Deprivation Therapy (ADT) (N=45)
Erectile disfunction (Reproductive system and breast disorders) | 4 (4) — Genitourinary AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT01517451/Prot_SAP_000.pdf